CLINICAL TRIAL: NCT04170101
Title: Randomized Controlled Trial Comparing the Impact of Deep Versus Moderate/Superficial NMB on Surgical Conditions and Muscle Trauma During Hip Arthroplasty by Direct Anterior Approach Using Minimally Invasive Surgery.
Brief Title: RCT Deep vs Moderat NMB on Surgical Conditions During THP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: AZ Sint-Jan AV (Other)
Responsible Party: Principal Investigator, Jan Mulier, Prof dr, AZ Sint-Jan AV
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2019RCTdeepNMBTHP
Record Dates: First submitted 2019-11-16; First posted 2019-11-20 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2020-03

CONDITIONS: Muscle Injury

STUDY DESIGN:
Intervention Model Description: a continuous deep NMB (group A) versus a non deep NMB (group B) having a moderate to superficial block imitating common practice today as control group.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- a continuous deep NMB (group A) (Experimental): after 0,6 mg/kg LBW Rocuronium for intubation Rocuronium is given in a continuous infusion starting at 1 mg/kg/h and adapted to keep PTC below 5 and note.
  Interventions: Procedure: deep NMB
- non deep NMB (group B) (Placebo Comparator): after 0,6 mg/kg LBW Rocuronium for intubation no extra NMB is given and depth is measured by TOF/PTC to note depth.
  Interventions: Procedure: moderate NMB

INTERVENTIONS:
Procedure: deep NMB — 0,6 mg/kg LBW Rocuronium is used to facilitate intubation, and followed by an infusion of 1 mg/kg LBW/h , further adapted to keep PTC < 3
  Arms: a continuous deep NMB (group A)
Procedure: moderate NMB — 0,6 mg/kg LBW rocuronium is used to facilitate intubation, not followed by an infusion or extra bolus.
  Arms: non deep NMB (group B)

SUMMARY:
A clinical deep NMB might relax the anterior muscles of the upper leg better than a moderate/superficial block giving a better exposure for the surgeon with less muscle trauma by traction to expose the hip.

a continuous deep NMB (group A) versus a non deep NMB (group B) having a moderate to superficial block imitating common practice today as control group.

Primary objectives are surgical exposure and Secondary objectives are Muscle damage creatine kinase changes, C-reactive protein (CRP), first time leaving bed postoperative, post operative pain as measured by opioid use postoperative at 24h, with a control of max VAS score during first 24 hour, length of hospital stay (LOS), number of adverse events using the Dindo-Clavien surgical complication score, QoR15 measured at 24h on the ward.

DETAILED DESCRIPTION:
In this study, CRP levels are choosen as it is measured standard in every total hip arthroplasty (THA) procedure. CK is a good biomarker for muscle trauma and therefore chosen as second marker.

The study is blinded for the treating surgeon, who will be making the assessment for the surgical conditions. The attending anesthesiologist is not blinded as he has to measure NMB in both groups and give a rocuronium infusion to stay deep in the study group. The anesthesiologist and the nurses following the patient on the post anesthetic care unit (PACU) and the ward are different from the attending anesthesiologist and are blinded. They will not be informed by the attending anesthesiologist on randomization allocation.

Randomization:

Group A deep NMB group:

• 0,6 mg/kg LBW Rocuronium is used to facilitate intubation, and followed by an infusion of 1 mg/kg LBW/h , further adapted to keep post tetanic count (PTC) < 3 without informing the surgeon of the depth (surgeon is blinded)

Group B moderate to superficial NMB group:

* 0,6 mg/kg LBW rocuronium is used to facilitate intubation, not followed by an infusion or extra bolus.train of four ( TOF) and PTC are measured at the beginning of surgery without informing the surgeon of the depth. (surgeon is blinded)

  2 weeks before surgery at consultation of orthopedics and anesthesia:
* Inclusion criteria, signing informed consent, CRP blood sample
* 15 Quality of recovery questions (QoR15) filled in to have a pre op status

Day before surgery:

* Verification that study can be performed ( equipment, surgeon, anesthesiologist and investigators available) Morning of surgery
* Control signing of informed consent is done and patient still willing to continue the study
* Attending anesthesiologist ask the randomization allocation at the secretary anesthesia without informing surgeon, colleagues and nurses on PACU and ward.

Anesthesia & surgery performed

* CRF is filled in with time stamps, dosing of drugs and monitoring values
* Surgeon is asked for a surgical exposure grading ( 1-5) after initial incision, at the critical moment of prosthesis insertion and before closure.
* In order to measure the degree of muscle damage, one light photo is taken of the muscles before closing and archived for later anonymous scoring by an independent orthopedic surgeon doing also THA by DAA but not around that day in the OR (3 surgeons do frequently THA by DAA).
* If an opioid is given before PACU admission dose and time are noted in the clinical registration file (CRF) PACU
* VAS score is recorded on admission, every hour and before leaving PACU.
* The total dose of opioids given during the PACU are noted in the CRF Ward
* Max visual analog pain score (VAS) during first 24 hours on the ward is noted in the CRF.
* The QoR15 is repeated at 24 hours post surgery
* A CRP blood sample is taken 24 hours post surgery
* The total dose of opioids given on the ward till discharge is noted in the CRF

Home

* 2 weeks after surgery a phone call is given to request healthy state
* and hear of any adverse event or complication.
* and repeat the QoR15 questionnaire by phone

ELIGIBILITY:
Inclusion Criteria:

* • Hip arthroplasty by anterior approach using Minimally Invasive Surgery

Exclusion Criteria:

* • Revision arthroplasty.

  * Allergy or contra indications to use any of the drugs included in anesthesia.
  * Addiction to or chronic opioid use before surgery.
  * Major cardiovascular, pulmonary, liver or renal insufficiency before surgery requiring possible post-operative intensive care admission.
  * Contra indication for a general anesthesia with intubation and mechanical ventilation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-04-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
surgical exposure | from incision till end of surgery stop at day zero
  After the surgical procedure the surgeon will be asked to score the surgical conditions on an adapted five point Leiden scale (validated scale):
  max = 5 and best; min = 1 and worst grade 5: optimal surgical conditions, perfect access to the hip joint and excellent visibility.
  grade 4: good conditions: adequate surgical conditions to perform the surgery, but not optimal grade 3: just acceptable conditions, surgical procedure is jeopardized, but adequate surgical result is still obtained, eventually after additional intervention grade 2: poor conditions, exposure and handling hindered resulting in suboptimal surgical outcome requiring adaptation of procedure or interventions to improve condition.
  grade 1: extremely poor conditions, the surgeon is unable to work because of the inability to get access to the hip joint because of inadequate muscle relaxation and request to improve conditions first before continuing.

SECONDARY OUTCOMES:
muscle injury | on photo after procedure stop at day zero
  This is scored on an adapted five point scale post surgery on a light photo taken at end of surgery before closing, by an orthopedic surgeon not around during surgery.
  max = 5 and best; min = 1 and worst
  grade 1: muscle severely damaged with open cuts; grade 2: muscle damaged with free tears; grade 3: muscle superficial damaged and swollen; grade 4: muscle intact, but swollen or perfusion not optimal grade 5: muscle intact without swelling and normal perfused.
creatinine kinase (CK) | 24 hours after surgery stop at day 1
  creatinine kinase (CK) changes as a measure for muscle trauma, at 24 hours postoperative versus baseline
C-reactive protein (CRP) | 24 hours after surgery stop at day 1
  C-reactive protein (CRP) changes as a measure for inflammation, at 24 hours postoperative versus baseline.
leaving bed | within 24 hours postoperative stop at day 1
  First time leaving bed postoperative
Length of stay | measured in days up to one week post surgery stop at day 7
  Length of hospital stay (LOS)
postoperative complications | up to two weeks postoperative stop at day 14
  Number of adverse events using the Dindo-Clavien surgical complication score
quality of recovery | 2 weeks postoperative stop at day 14
  15 Quality of recovery questions (QoR15) measured at 24h on the ward and at 2 weeks post operative max: 150: best; min: 0: worst each question is answered on a scale from 0 to 10.

CONTACTS AND LOCATIONS:
Overall Officials: jan mulier, Principal Investigator — AZSint Jan AV
Locations (1):
- Azsintjan, Bruges, Belgium

IPD SHARING:
Plan to Share IPD: No